CLINICAL TRIAL: NCT02941887
Title: Down's Syndrome Patients Behavior Correlations to Periodontal Disease Status
Brief Title: Global Behavior and Periodontal Disease in Down's Syndrome Patients
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Carla Andreotti Damante, Associate professor, University of Sao Paulo
Other Study IDs: FOBDownSyndrome2
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Behavior; Periodontal Diseases
Keywords: Social behavior; Gingivitis; Periodontitis; Down's Syndrome
MeSH Terms: conditions — Behavior; Periodontal Diseases; Social Behavior; Gingivitis; Periodontitis; Down Syndrome | interventions — Applied Behavior Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Down's Syndrome: Behavior analysis in Down's Syndrome patients
  Interventions: Behavioral: Behavior Analysis

INTERVENTIONS:
Behavioral: Behavior Analysis — One examiner observed global behavior of patients during a dental care session, guided by a behavioral scale.

SUMMARY:
This study aimed at correlating global behavior of Down's Syndrome patients to periodontal disease status.

DETAILED DESCRIPTION:
There is a higher prevalence and severity of periodontal disease in Down's Syndrome patients. Plaque levels in these patients are high due to poor hygiene habits. Behavior also may contribute to the overall periodontal condition.

ELIGIBILITY:
Inclusion Criteria:

* Down's Syndrome Diagnose characterized by the whole chromosomal aneuploidy 15 to 52 years
* Absence of severe hearing loss could impair the comprehension about the dental treatment
* Absence of severe visual loss that could impair the comprehension about the dental treatment
* Presence of at least four teeth being one for hemiarch.
* Diagnose of gingivitis and periodontitis
* Absence of acute periodontal disease and necrotizing periodontal disease.

Exclusion Criteria:

* Smokers
* Use of alcohol
* Menopause
* Pregnancy
* Absence of all teeth
* Uncontrolled diabetes mellitus
* Uncontrolled hyperthyroidism
* Angina
* Uncontrolled hypertension
* Coagulopathy
* Use of illicit drugs
* Head and neck radiotherapy
* Chemotherapy
* Non-cooperative patients or patients with other diseases as autism.

Ages: 15 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with a medical diagnose of Down's Syndrome
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Periodontal disease (gingivitis and periodontitis) measured by a periodontal probe and classified according to severity | One day
  Severe periodontitis was defined by the presence of ≥ 2 interproximal sites in different teeth with clinical attachment level (CAL) ≥ 6mm and ≥1 interproximal site with pocket probing depth (PPD) ≥5mm. Moderate periodontitis was defined by the presence of ≥ 2 interproximal sites in different teeth with CAL ≥ 4mm or ≥ 2 interproximal sites in different teeth with PPD ≥5mm. Mild periodontitis was defined as ≥ 2 interproximal sites in different teeth with ≥ 3 mm CAL and ≥ 2 interproximal sites in different teeth with ≥ 4 mm PPD or at least 1 site with PPD ≥ 5 mm (20,21). Gingivitis was determined as follows: Subjects were considered healthy if presented PPD ≤3mm/BOP extent scores < 10% and with gingivitis if presented PPD ≤3mm/ bleeding on probing (BOP) extent scores >10%. Prevalence of periodontal disease was the sum of gingivitis, mild, moderate and severe periodontitis.
Global behavior - observation and scoring based on a behavior scale | One day
  Behavioral aspects: Interaction to evaluator, Communicative intention, Attention time, Response to conversation, Comprehension of concrete/no concrete situations with/without visual support, Parental interference, Acceptance of activities, Mimic, Eye contact, Participation in the dialogue (speech), Logical time sequence, Dialogue keeping, Word production
  Scores: 0 - absence, 1 - strictly presented, 2 - evidently presented.

CONTACTS AND LOCATIONS:
Locations (1):
- Bauru School of Dentistry, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Startin CM, Rodger E, Fodor-Wynne L, Hamburg S, Strydom A. Developing an Informant Questionnaire for Cognitive Abilities in Down Syndrome: The Cognitive Scale for Down Syndrome (CS-DS). PLoS One. 2016 May 6;11(5):e0154596. doi: 10.1371/journal.pone.0154596. eCollection 2016. PMID 27153191